CLINICAL TRIAL: NCT05696886
Title: The Effect of Intraoperative Tramadol on Postoperative Opioid Requirements After Laparoscopic Sleeve Gastrectomy for Morbid Obese Patients (A Retrospective Multicentric Cohort Study)
Brief Title: The Effect of Intraoperative Tramadol on Postoperative Opioid
Acronym: LSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Clinical Professor, Gastroenterology surgical center, mansoura university, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.23.01.2008
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain
Keywords: laparoscopic sleeve gastrectomy; morbid obesity; postoperative pain; tramadol; pethidine
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid | interventions — Meperidine; Tramadol

STUDY DESIGN:
Intervention Model Description: Group A received Pethidine alone in the period between January 2021 and December 2021, while Group B got Tramadol with pethidine in the period between January 2022 and December 2022. Doses were based on the patient's actual body weight.
Who Masked: Participant
Masking Description: Group A received Pethidine alone in the period between January 2021 and December 2021, while Group B got Tramadol with pethidine in the period between January 2022 and December 2022. Doses were based on the patient's actual body weight.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A received Pethidine alone in the period between January 2021 and December 2021, (Active Comparator): received Pethidine alone in the period between January 2021 and December 2021, while
  Interventions: Drug: Pethidine
- Group B got Tramadol with pethidine in the period between January 2022 and December 2022. (Active Comparator): Group B got Tramadol with pethidine in the period between January 2022 and December 2022.
  Interventions: Drug: Tramadol with pethidine

INTERVENTIONS:
Drug: Pethidine — Group A received Pethidine alone in the period between January 2021 and December 2021
  Other Names: Group A
  Arms: Group A received Pethidine alone in the period between January 2021 and December 2021,
Drug: Tramadol with pethidine — Group B got Tramadol with pethidine in the period between January 2022 and December 2022
  Other Names: Group B
  Arms: Group B got Tramadol with pethidine in the period between January 2022 and December 2022.

SUMMARY:
Postoperative pain remains a very UNPLEASENTevent, particularly in morbidly obese patients that may be associated with obstructive sleep apnea. Bariatric surgery patients must get safe and efficient analgesia, which is essential given that up to 45 % of patients report substantial pain in the first two days following surgery. The study's purpose was to compare the efficacy and safety of combined tramadol with pethidine versus pethidine alone and to assess their impact on postoperative pethidine requirements after LSG for morbidly obese patients

DETAILED DESCRIPTION:
This multicenter cohort research included patients with morbid obesity who had LSG between January 2021 and December 2022. The patients included in the study were allocated to one of two treatment groups that were not randomized but the patients were categorized according to the time of surgery: Group A received Pethidine alone in the period between January 2021 and December 2021, while Group B got Tramadol with pethidine in the period between January 2022 and December 2022. Doses were based on the patient's actual body weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients with morbid obesity defined as a BMI of more than 40 or
* BMI less than 35 with at least one comorbidity and
* ages ranging from 16 to 65, were patients

Exclusion Criteria:

* Patients under the age of 16 or over 65,
* Those with severe GERD, leakage
* pregnancy, or
* inflammatory bowel disease,

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — 16-65
Enrollment: 400 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
VAS of pain | 48 hours postoperative
  the severity of pain
opioid requirement | one month
  the need of pethidine

SECONDARY OUTCOMES:
hospital stay | one month
  hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ayman E Nakeeb, Principal Investigator — Mansoura University, Gastrointestinal Surgery Center
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Outside U.S and Canada, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the study protocol will be available for another researcher
Supporting Information: Study Protocol
Time Frame: available for any researcher at any time
Access Criteria: elnakeebayman@yahoo.com
URL: http://www.mans.edu.eg/

REFERENCES:
- [Result] Zeeni C, Aouad MT, Daou D, Naji S, Jabbour-Khoury S, Alami RS, Safadi BY, Siddik-Sayyid SM. The Effect of Intraoperative Dexmedetomidine Versus Morphine on Postoperative Morphine Requirements After Laparoscopic Bariatric Surgery. Obes Surg. 2019 Dec;29(12):3800-3808. doi: 10.1007/s11695-019-04074-1. PMID 31286397
- [Result] Zhang Y, Zhou Y, Hu T, Tong X, He Y, Li X, Huang L, Fu Q. Dexmedetomidine reduces postoperative pain and speeds recovery after bariatric surgery: a meta-analysis of randomized controlled trials. Surg Obes Relat Dis. 2022 Jun;18(6):846-853. doi: 10.1016/j.soard.2022.03.002. Epub 2022 Mar 9. PMID 35422388
- [Result] Tian C, Lee Y, Oparin Y, Hong D, Shanthanna H. Benefits of Transversus Abdominis Plane Block on Postoperative Analgesia after Bariatric Surgery: A Systematic Review and Meta-Analysis. Pain Physician. 2021 Aug;24(5):345-358. PMID 34323436
- See also: mansoura university — http://www.mans.edu.eg/